CLINICAL TRIAL: NCT03753555
Title: The Effect of InTensive Statin in Ischemic Stroke With inTracranial Atherosclerotic Plaques: a Prospective, Random, Single-center Study Based on High Resolution Magnetic Resonance Imaging
Brief Title: The Effect of InTensive Statin in Ischemic Stroke With inTracranial Atherosclerotic Plaques
Acronym: INSIST-HRMRI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Department Chairman, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k（2018）44
Record Dates: First submitted 2018-11-13; First posted 2018-11-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Atherosclerosis, Cerebral
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis | interventions — Atorvastatin; Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine-dose statin group (Active Comparator): Routine-dose statin group will be gaven the treatment of atorvastatin 20mg Qd for 12 months
  Interventions: Drug: Atorvastatin Calcium
- high-dose statin or PCSK9 inhibitor group (Experimental): high-dose statin group will be gaven the treatment of atorvastatin 40-80mg Qd till 6 months at the moment the subjects will be followed up to determine plaques status by HRMRI examination, among which the subjects presenting culprit plaque progression with the significant increasing of plaque burden including intraplaque hemorrhage will be again randomized into two groups at a ratio of 1:1 as followed: atorvastatin-probucol group will be administrated atorvastatin 40-80mg Qd plus probucol 0.5g Bid till 12 months, the other group will maintain the original scheme till 12 months.
  PCSK9 inhibitor group will receive the subcutaneous injection of Evolocumab (140mg, 2 / month) for one year.
  Interventions: Drug: Atorvastatin Calcium; Drug: Probucol; Drug: PCSK9 inhibitor

INTERVENTIONS:
Drug: Atorvastatin Calcium — 20mg Qd for 12 months
  Arms: Routine-dose statin group
Drug: Atorvastatin Calcium — 40-80mg Qd for 6 months
  Arms: high-dose statin or PCSK9 inhibitor group
Drug: Probucol — 0.5g Bid for 6 months
  Arms: high-dose statin or PCSK9 inhibitor group
Drug: PCSK9 inhibitor — Evolocumab 140mg subcutaneously injected, twice each month
  Arms: high-dose statin or PCSK9 inhibitor group

SUMMARY:
Intracranial atherosclerotic disease is the most common cause of ischemic stroke that is directly attributed to the progression or rupture of intracranial high-risk plaque in Asia. Many studies mainly from Euro-American population with a focus on extracranial carotid plaque have fully demonstrated the advantages of intensive statin therapy on stabilizing or reversing plaque burden, reversing plaque composition presenting that lipid-rich necrotic core (LRNC) is gradually replaced by fibrous tissue, and even reversing pattern of arterial remodeling to reduce the occurrence of cerebrovascular events. Yet, direct evidence of the effect of intensive statin therapy on intracranial atherosclerotic plaques is lacking and the effect of statin intensity and duration on intracranial plaque burden and composition is still unclear. High resolution magnetic resonance imaging (HRMRI) is a new and non-invasive technique that enable to assess the morphologic characteristics of vascular wall and plaque composition of intracranial artery. Based on above discussion, the investigators conduct this study to further determine the effect of intensive statin in ischemic stroke with intracranial atherosclerotic plaques.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18-80 years
2. Time of onset: within 1 week
3. NIHSS score ≤12
4. Acute ischemic stroke confirmed by head CT or MRI
5. Premorbid mRS ≤1
6. The degree of stenosis of carotid artery, vertebral artery and intracranial portion of internal carotid artery on the lesion side <50%
7. The culprit plaque or possible culprit plaque with plaque burden of 40% or more found by HRMRI in the proximal part of the middle cerebral artery M1 segment or basilar artery of ipsilateral lesion
8. Signed informed consent

Exclusion Criteria:

1. Intracranial hemorrhage found by head CT
2. Stroke attributable to cardioembolic origin (atrial fibrillation, valvular heart disease, aortic arch atherosclerosis)
3. Severe hepatic or renal dysfunction
4. Pregnant females
5. Abnormal elevation of creatine phosphokinase
6. Expected stent angioplasty
7. Blood sugar is out of control
8. Receiving statins within 1 month before onset
9. Obstinate hypertension with more than 140/90 mmHg after medication
10. Not willing and able to comply with scheduled visits, lifestyle guidelines, treatment plan, laboratory tests, and other study procedures
11. Unsuitable for this clinical studies assessed by researcher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in remodeling index after the statin treatment | baseline, 6 months, 12 months after treatment
  remodeling index: crimed vessel area/normal vessel area on high-resolution MRI
Changes in plaque burden after the statin treatment | baseline, 6 months, 12 months after treatment
  plaque burden: crimed vessel wall area/crimed vessel area on high-resolution MRI
Changes plaque composition in after the statin treatment | baseline, 6 months, 12 months after treatment
  plaque composition: lipid core and fiber tissue of plaque on high-resolution MRI

SECONDARY OUTCOMES:
level of serum bio-markers compared with baseline | 6 months
  Serum level of LDL、hs-CRP、sLOX1 and oxLDL
level of serum bio-markers compared with baseline | 12 months
  Serum level of LDL、hs-CRP、sLOX1 and oxLDL
mRS (0-2) | 6 months
  proportion of mRS (0-2)
mRS (0-2) | 12 months
  proportion of mRS (0-2)
vascular events | 6 months
  incidence of Transient ischemic attack, stroke or other vascular events
vascular events | 12 months
  incidence of Transient ischemic attack, stroke or other vascular events
abnormal test data | 12 months
  incidence of abnormal liver function or muscle enzyme levels
any adverse event | 12 months
  incidence of adverse event
death of any causes | 12months
  proportion of death

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China